CLINICAL TRIAL: NCT01596192
Title: The Sensitivity and Specificity of 18F-Fluorodeoxyglucose Positron Emission Tomography -Computed Tomography for the Diagnosis and Monitoring of Acute Graft vs. Host Disease
Brief Title: PETCT for Diagnosing and Monitoring Acute GVHD
Acronym: PETGVHD-001
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RMC-PETGVHD-001
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-02

CONDITIONS: Acute Graft Versus Host Disease
Keywords: allogeneic transplantation, GVHD; Patients with acute GVHD after allogeneic hematopoietic cell transplantation
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Levels of HGF, IL8, IL2R and TNFR1 will be measured at the onset of GVHD and prior to the second PET-CT. Five cc blood will be drawn twice from each patient and will be collected in an EDTA containing tube.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with acute GVHD: Patients after allogeneic hematopoietic cell transplantation who have developed acute GVHD
  Interventions: Other: PETCT

INTERVENTIONS:
Other: PETCT — CT-PET will be performed within 3 days from acute GVHD diagnosis. Each patient will receive 400-610 MBq (11-16.5 mCi) of 18F-FDG intravenously. After tracer injection, the patients will rest on a comfortable chair during the 18F-FDG-uptake period, and drink with 150-300mg Levolac (Fresenius Kabi, Austria) diluted in 1000-1500cc water. CT-PET will be initiated 45-50 min after injection of the 18F-FDG.ll scans will be performed on a Discovery STE PET/CT scanner (General Electric Medical Systems, Milwaukee, WI).
  CT will be performed 45-50 minutes after drinking the diluted lactulose solution had been ingested. The CT images will be acquired from the diaphragm to the symphysis pubis. After IV administration of 100 ml of nonionic contrast medium at a flow rate of 2.5 ml/sec.

SUMMARY:
Graft versus host disease (GVHD) is one of the major causes of death in patients undergoing allogeneic hematopoietic cell transplantation. 18F-FDG PET/CT (2-[fluorine-18] fluoro-2-deoxy-D-glucose, Positron emission tomography- CT) is a noninvasive technique that allows quantifying and precisely localizing 18F-FDG uptake in the entire body. 18F-FDG uptake is caused by increased local metabolic activity. In this study, we aim to evaluate and characterize the correlation between CT-PET findings in patients suspected to have acute GVHD, and the disease course.

DETAILED DESCRIPTION:
Graft versus host disease (GVHD) is one of the major causes of death in patients undergoing allogeneic hematopoietic cell transplantation (HCT). Despite prophylactic measures, the incidence of acute GVHD is estimated at 40-60% among patients receiving allograft from HLA-identical sibling donors, and may even reach 75% in patients receiving HLA-matched unrelated grafts. Approximately 20% of the patients will develop the severe variant of the disease and there is a tight association between the severity of GVHD and transplantation-related-mortality. The treatment of GVHD is largely based on high dose steroids regimen which is associated with long term morbidity and mortality. In the subgroup of patients with steroid-refractory or slowly resolving GVHD, there are currently no recommendations on the best timing of tapering down the steroids dose in the case of resolution of the disease, or adding a second line medication, in case of non-resolving or progression of the symptoms.

18F-FDG PET/CT (2-[fluorine-18] fluoro-2-deoxy-D-glucose, Positron emission tomography- CT) is a noninvasive technique that allows quantifying and precisely localizing 18F-FDG uptake in the entire body. 18F-FDG uptake is caused by increased local metabolic activity. Such increased uptake has been described not only in neoplastic lesions but also in inflammatory lesions (2). In this condition, uptake has been correlated with local stimulation of tumor necrosis factor, and with monocyte priming and activation. A physiologic variable uptake may be observed in the bowel, especially the cecum, and has limited the use of PET in inflammatory bowel diseases. The advantage of combined PET and CT devices leads to significant improvements in the interpretation of the bowel areas, and greatly reduces the number of false-positive findings in the gastrointestinal tract.

CT-PET has been recently evaluated in our center as a diagnostic tool for Crohn disease. In this study, CT-PET had a good correlation between FDG uptake and the severity of Crohn disease. In the acute GVHD setting, a study reported on a small cohort suggested a correlation between CT-PET findings, FDG uptake, and the diagnosis of lower gut acute GVHD.

In this study, we aim to evaluate and characterize the correlation between CT-PET findings in patients suspected to have acute GVHD, and the disease course.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with grade 2-4 acute GVHD
2. Age> 18 years
3. Signing an informed consent

Exclusion Criteria:

1. Men or women less than 18 years of age
2. Severe Hyperglycemia (>500 mg/dL)
3. Severe allergy to iodine contrast
4. Extremely sick patients who cannot be transported to the PET unit
5. Unable to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the BMT unit, Beilinson Hospital with the diagsnosis of acute GVHD
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Change of gut FDG uptake at onset and after treatment with steroids in patients with acute GVHD | At the onset of GVHD (up-to 6 months after hematopoietic cell transplantation) and then after 4 weeks from the date of first CT-PET (up-to 7 months after transplantation)
  CT-PET will be performed at the onset of GVHD(up-to 6 months from transplantation) and repeated after 4 weeks. The findings will be compared with the initial CT-PET results. The time frame of 4 weeks is the period of time in which most patients become either asymptomatic or in need for additional immunosuppressive therapy. In addition, all patients will go through the standard GVHD evaluation practice which includes (but not limited to) GI endoscopy (sigmoidoscopy and/or gastroscopy) and skin biopsies. Data obtained from the CT PET results will be compared with the GI findings.

SECONDARY OUTCOMES:
Correlation between blood cytokines level and PETCT results | At the onset of GVHD (up-tp 6 months post transplantation) and then, after 4 weeks (up-to 7 months from transplantation)
  Levels of HGF, IL8, IL2R and TNFR1 will be measured at the onset of GVHD and prior to the second PET-CT. Five cc blood will be drawn twice from each patient and will be collected in an EDTA containing tube. Cytokines levels will be measured as previously described

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ram, M.D., Principal Investigator — BMT Unit, Davidoff Cancer Center, Rabin Medical Center, Beilinson Hospital
Locations (1):
- BMT unit, Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel